CLINICAL TRIAL: NCT05476536
Title: The Effectiveness of Technology Combined Self-health Management and Home Care Model Improved the Metabolic Diseases, Sarcopenia, and Serum Inflammation and Metabolic Markers Among Middle-aged and Elderly Individuals in the Community
Brief Title: Effectiveness of Technology for Metabolic Diseases Combined Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung University of Science and Technology (Other)
Collaborators: Chang Gung Memorial Hospital (Other); Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Shu-Hung Chang, Professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MOST-110-2314-B-255-007-
Record Dates: First submitted 2022-07-19; First posted 2022-07-27 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Metabolic Disease
Keywords: self-health management; metabolic diseases; sarcopenia; frailty; intervention
MeSH Terms: conditions — Metabolic Diseases; Sarcopenia; Frailty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): self-management skills and healthy technology APP
  Interventions: Behavioral: self-management skills and healthy technology APP
- control group (No Intervention): Health education leaflet

INTERVENTIONS:
Behavioral: self-management skills and healthy technology APP — self-management skills and healthy technology APP
  Arms: experimental arm

SUMMARY:
The lifestyle program intervention program focusing on healthy dietary habit and exercise effectively prevents metabolic syndrome, sarcopenia or frailty. Thus, the purpose of this study was to assess the efficacy of intervention program on metabolic syndrome subjects in Taiwan.

DETAILED DESCRIPTION:
The study is a 2-parallel groups' randomized controlled trial. Participants with metabolic syndrome (three or more risk factors - triglycerides (TG) >150 mg/dL, systolic blood pressure (SBP) ≥130 mm Hg, diastolic blood pressure (DBP) ≥85 mm Hg, or fasting blood glucose≥100 mg/dL; high-density lipoprotein cholesterol<50 mg/dL, or waist circumference ≥80 cm) are enrolled. The four community units are randomized to receive a lifestyle intervention (intervention arm) or an education leaflet (control arm). The parameters are obtained from physical examination and biochemical assessments by well-trained case manager at baseline and 4th months. All participants complete a structured questionnaire, including basic information, SOF, physical performance, physical activity, and food-frequency.

ELIGIBILITY:
Inclusion Criteria:

* older adult with age ≥ 40 years
* community-dwelling
* no hearing and visual acuity difficulties

Exclusion Criteria:

* Unconscious
* Cognitive impairment or dementia

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
metabolic syndrome | 4 month follow up
  changes in triglycerides, high-density lipoprotein cholesterol, systolic blood pressure, diastolic blood pressure, fasting blood glucose, waist circumference
body weight | 4 month follow up
  weight in kilograms
BMI | 4 month follow up
  weight and height will be combined to report BMI in kg/m^2
Frailty | 4 month follow up
  measurement used study of osteoporotic fracture index (SOF).

SECONDARY OUTCOMES:
short physical performance battery | 4 month follow up
  sit-to-stand, standing balance, and gait-speed
upper limb muscle strength | 4 month follow up
  hand-grip strength
static balance ability | 4 month follow up
  single-leg standing with the eyes open
physical agility and dynamic balance ability | 4 month follow up
  Timed-Up and Go and Functional Reach Test

OTHER OUTCOMES:
Physical activity | 4 month follow up
  used International Physical Activity Questionnaire (IPAQ)
dietary behaviors | 4 month follow up
  intake rate of whole grains, vegetables, fruits, proteins, dairy products, and nuts.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hung Chang, Ph.D, Principal Investigator — Chang Gung University of Science and Technology
Locations (1):
- Taoyuan, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No